CLINICAL TRIAL: NCT00812630
Title: A Two-part Trial Assessing the Effects of 7α-methyl-19-nortestosterone (MENT) on Blood Pressure in Normal Men: an Open-label Pilot Study Followed by a Randomized, Double-blind, Placebo-controlled Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Population Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: Population Council #412
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Blood Pressure
Keywords: male hormonal contraception; Blood pressure, sperm concentration
MeSH Terms: interventions — trestolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): In the second part of the trial, subjects will apply MENT or placebo gel transdermally for 12 weeks and will have 24-hour blood pressure monitoring at baseline, Week 6 and Week 12.
  Interventions: Drug: MENT or placebo

INTERVENTIONS:
Drug: MENT or placebo — A dose of 1600µg/d of MENT will be delivered daily using a gel formulation containing 8.0 mg of MENT per 1.0 mL (delivering 800µg/d). Two mLs of gel will be applied daily for four weeks in the pilot study (by 6 men) and for 12 weeks in the main trial (by 62 men).

SUMMARY:
This is a two-part trial assessing the effects of MENT on blood pressure. The first part of the trial is an open-label pilot study to verify the MENT gel formulation delivers appropriate drug levels. Upon confirming MENT serum levels are within the required range, clinical trial material will be produced and labeled. Consequently, the second part of the trial, the main study, will proceed approximately two months after the conclusion of the pilot study. The main study, is a randomized, double-blind, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men age 18-40
* Man has a sperm concentration of greater than or equal to 15 x 106/mL at screening
* Man has not used hormonal therapy in the last six months
* Man has a testosterone level between 270-1070 ng/dL at screening

Exclusion Criteria:

* Man is hypertensive, defined by
* diastolic BP greater than or equal to 85 mmHg or systolic BP greater than or equal to 140 mmHg (the average of the 2nd and 3rd of 3 measurements after 10 minutes rest) at screening or
* a baseline ABPM average of diastolic greater than or equal to 85 mmHg systolic greater than or equal to 130 mmHg or
* is taking any hypertensive medication
* Man has a BMI over 33 kg/m2
* Man has active or a history of cerebrovascular or cardiovascular disease
* Man has chronic or acute liver or renal disease
* Man has a history of a significant psychiatric disorder, including severe depression
* Man has dermatitis, psoriasis or other severe skin disorder
* Man has clinically significant abnormalities of laboratory safety tests

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2008-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To assess the effects of MENT gel on blood pressure as compared to placebo gel. | 4 weeks

SECONDARY OUTCOMES:
To evaluate the serum levels of MENT, testosterone, DHT, LH, FSH and estradiol and their variation under therapy | 4 weeks
To assess the effects of MENT on sperm concentration | 21 months
To evaluate the safety and tolerability of MENT. | 21 months

CONTACTS AND LOCATIONS:
Overall Officials: Regine Sitruk-Ware, MD, Study Director — Population Council
Locations (1):
- The New York Presbyterian Hospital-Weill Cornell Medical Center, New York, New York, United States